CLINICAL TRIAL: NCT02511028
Title: In Vivo Characterization of Inflammation With Ferumoxytol, an Ultrasmall Superparamagnetic Iron Oxide Nanoparticle, on 7 Tesla Magnetic Resonance Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 150156; 15-N-0156
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-17

CONDITIONS: Multiple Sclerosis
Keywords: MRI; Multiple Sclerosis; Healthy Volunteer
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ferumoxytol (Experimental): A 510 mg dose (17 mL) of ferumoxytol diluted in 50 mL of 0.9% normal saline will be intravenously infused over 17 minutes
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — 510mg (17mL) IV

SUMMARY:
Background:

- Contrast agents help things show up better on magnetic resonance imaging (MRI) scans. Researchers want to see if the drug ferumoxytol is a good contrast agent. They want to determine that it does not cause prolonged MRI changes in the brain and to see if it helps identify inflammation in multiple sclerosis

Objective:

- To learn how ferumoxytol can be used to image inflammation in multiple sclerosis (MS).

Eligibility:

* Adults ages 18 70 who have MS.
* Healthy volunteers ages 18 70.

Design:

* Participants will have 5 clinic visits over 6 months.
* Participants will be screened with a medical history, neurological exam, and blood draw. Full clinical measures will be obtained.
* Participants will have a 7 tesla brain MRI scan that may include gadolinium contrast agent. The MRI is a metal cylinder in a strong magnetic field. The participant will lie on a table that can slide in and out of the cylinder.
* During visit 2, ferumoxytol with be given through a catheter (a thin plastic tube) that is inserted with a needle into a vessel in the arm.

<TAB>- Participants will then have a 7 tesla MRI scan of the brain..

* At each of the next 3 clinic visits, participants will have a 7 tesla brain MRI and have blood drawn. The MRIs may include gadolinium.
* Participants may have a full neurologic exam at these visits. At the final visit, full clinical measures will be obtained.
* Participants may have more MRI scans if a 6-month MRI shows ferumoxytol still in the brain.

DETAILED DESCRIPTION:
Objective

The goals of this pilot study are to (1) demonstrate the safety of ferumoxytol, a United States Food and Drug Administration (FDA) approved drug used in the treatment of iron deficiency anemia, as a contrast agent for brain magnetic resonance imaging (MRI), as determined by a lack of long-term signal change in healthy volunteers (HV) and people with multiple sclerosis (MS); (2) determine if ferumoxytol enhancement can be detected in MS lesions on 7-tesla (T) MRI; and (3) examine the spatial and temporal enhancement patterns of ferumoxytol compared to patterns seen with gradient-echo imaging and gadolinium contrast in MS lesions.

Study population

Up to 10 HVs and up to 10 participants with MS will be recruited for this study.

Design

Participants will undergo a series of brain MRIs on a 7 T scanner. MRI will be before (baseline) and 0-8 hours, 24-96 hours, 1 month, and 6 months following ferumoxytol administration.

Outcome measures

The primary outcome measure is change in gradient-echo T2-weighted signal (derived from an MR sequence sensitive to paramagnetic agents such as iron) in the globus pallidus, a known brain iron reservoir, 6 months following ferumoxytol administration. Thus, we will determine if ferumoxytol induces long-lasting brain signal intensity changes in HV and MS. Secondary outcome measures are: (1) the number, location, and qualitative morphology of ferumoxytol, gradient-echo phase, and gadolinium-enhanced MS lesions and how these lesions change over time; and (2) quantitative estimates of change in iron concentration by determining R2 (= 1/T2) relaxation rate within MS lesions, normal appearing white matter, normal appearing gray matter, and other iron-rich regions within the brain before and after ferumoxytol injection.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY VOLUNTEER INCLUSION CRITERIA

* age between 18 and 70 (inclusive)
* able to give informed consent
* brain MRI within 2 years of study enrollment that shows no clinically significant abnormalities, in the judgment of a board-certified and NIH-credentialed neuroradiologist

PATIENT INCLUSION CRITERIA

* age between 18 and 70, inclusive
* able to give informed consent
* diagnosis of multiple sclerosis according to revised McDonald Criteria

EXCLUSION CRITERIA:

GENERAL EXCLUSION CRITERIA:

* screening labs demonstrating any value for hepatic or renal function levels out of the range of normal, to include AST, ALT, bilirubin, alkaline phosphatase, creatinine, eGFR
* evidence of polycythemia vera with hemoglobin levels more than 1 standard deviation above the NIH laboratory s normal level
* iron overload syndromes, including hemochromatosis, or subjects with evidence of iron overload with a baseline ferritin level greater than 370 ng/ml and percent saturation of transferrin level greater than 40%.
* previous or current alcohol and/or substance abuse per medical history or medical records
* medical contraindications for MRI (e.g., any non-organic implant or other device such as a cardiac pacemaker or infusion pump or other metallic implants, objects, or body piercings that are not MRI-compatible or cannot be removed)
* psychological contraindications for MRI (e.g., claustrophobia), to be assessed at the time the medical history is collected
* pregnancy or current breastfeeding
* reported history of clinically significant impaired hearing, because people with impaired hearing are at increased risk of sound-induced damage from the MRI scanner
* known allergy to dextran or drugs containing iron salts or any previous history of severe allergic reactions, anaphylaxis, to any drug
* clinically significant medical or neurological disorders that, in the judgment of the investigators might expose the patient to undue risk of harm confound study outcomes or prevent the participant from completing the study; examples of such conditions include but are not limited to diagnosis of certain types of cancer, cardiopulmonary conditions such as congestive heart failure, or uncontrolled hypertension

ADDITIONAL PATIENT EXCLUSION CRITERION:

-4 or more gadolinium-enhancing lesions on the screening scan

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
change in gradient-echo T2*-weighted signal in an iron-rich brain structure, the globus pallidus | 6 months following ferumoxytol administration
  determine if ferumoxytol induces long-lasting brain signal intensity changes in HV and MS

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-N-0156.html